CLINICAL TRIAL: NCT00055588
Title: Spinal Substrates of Training-Dependent Improvements in Locomotor Function
Brief Title: Nervous System Function in Normal Volunteers During Cycling Training
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030120; 03-N-0120
Record Dates: First submitted 2003-03-06; First posted 2003-03-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-05-20

CONDITIONS: Healthy
Keywords: Spinal Reflexes; Motor Practice; Spinal Cord Injury; Locomotion; Healthy Volunteer; HV
MeSH Terms: conditions — Spinal Cord Injuries

INTERVENTIONS:
Procedure: Locomotor training

SUMMARY:
This study will identify changes that occur in the nervous system of healthy normal volunteers while they are learning a cycling task.

Healthy subjects 18 years of age and older who can cycle for 16 minutes may be eligible for this study. Candidates will be screened with a brief medical history and physical examination.

Participants will be assigned to one of three groups:

* Complex training: Cycling for 16 minutes at a constant speed of 60 rpm with frequent changes in pedal resistance.
* Simple training: Cycling for 16 minutes at a constant speed of 60 rpm with no changes in pedal resistance.
* No training: Remaining seated on the bike for 16 minutes performing no exercise.

Participants will cycle for 16 minutes for the training task, plus 4 minutes before and after the training. Reflexes will be measured with nerve conduction studies and somatosensory evoked potential (SSEP) recordings before and after training. Nerve conduction studies measure the speed with which nerves conduct electrical impulses and the strength of the connection between the nerve and the muscle. For these studies, a probe is placed on the skin over the calf muscles and the knee to deliver a small electrical stimulus, and wires are taped to the skin to record the impulses. SSEP recordings, which measure of the excitability of the brain to sensory stimuli, are collected from electrodes placed on the scalp.

After the training period, multiple train stimulation (MTS) is applied for 10 minutes. For MTS, weak electrical currents are delivered for 10 seconds every 10 seconds. These stimuli produce a buzzing sensation without pain, discomfort, or muscle twitching. The MTS is followed by another 4 minutes of cycling.

Participants also undergo transcranial magnetic stimulation (TMS). For this procedure, an insulated wire coil is held over the scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that travels through the scalp and skull and causes small electrical currents in the brain cortex (outer part of the brain). The stimulation may cause twitching in the muscles of the face, arm, or leg. The electrical activity of the muscles is recorded with a computer or other recording device, using electrodes attached to the skin with tape.

DETAILED DESCRIPTION:
In a previous study, we have shown that locomotor training with frequent changes in pedal resistances (complex training) elicits significant improvement in locomotor performance compared to training consisting of constant pedal resistance (simple training). Behavior gains associated with complex training correlate with down-regulation in the excitability of the alpha-motoneurone pools controlling muscles involved in the training task, as measured by changes in the soleus H-reflex, raising the hypothesis of a cause-effect link between performance improvements and modulation of spinal cord function. The purpose of this protocol is to determine if down-regulation in the excitability of the alpha-motoneuron pool is required for the improvement in locomotor performance. To address this issue, we hypothesize that up-regulation of alpha-motoneuron excitability will cancel improvements in locomotor performance elicited by complex training more than in subjects undergoing a period of simple training. The results of this study would provide novel information on the spinal substrates underlying learning of a locomotor task in intact humans and could be relevant to the design of rehabilitative strategies in patients with locomotor disorders.

ELIGIBILITY:
* INCLUSION CRITERIA:

Normal volunteers (ages 18 and above) who are willing to participate and who are considered able to cycle for16 minutes based on neurological and physical exams.

EXCLUSION CRITERIA:

1. Subjects with history of heart condition, unresponsive arterial hypertension, diabetes, chronic back pain, sciatica, peripheral neuropathy, rheumatoid arthritis, active joint deformity of arthritic origin, alcohol or drug abuse, psychiatric disorder requiring hospitalization or prolonged treatment, head injury with loss of consciousness, epilepsy.
2. Subjects with cardiac pace-makers, intracardiac lines, or implanted medication pumps.
3. Subjects with history of hyperthyroidism or individuals receiving drugs acting primarily on the central nervous system or disorders of the blood coagulation system.
4. Subjects with eye, blood vessel, cochlear, or eye implants.
5. Subjects with increased intracranial pressure as evaluated by clinical means.
6. Subjects with metal in the cranium except in the mouth.
7. Subjects with metal fragments from occupational exposure or surgical clips in or near the brain.
8. Women in the last trimester of pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-03-04; Study Completion 2008-05-20

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Boroojerdi B, Ziemann U, Chen R, Butefisch CM, Cohen LG. Mechanisms underlying human motor system plasticity. Muscle Nerve. 2001 May;24(5):602-13. doi: 10.1002/mus.1045. PMID 11317269